CLINICAL TRIAL: NCT04978597
Title: A Phase III, Double-Blind, Randomized, Placebo-Controlled and Parallel-Group Study to Evaluate the Efficacy and Safety of Opicapone, as Add-on to Stable Levodopa (L-DOPA) Plus a Dopa Decarboxylase Inhibitor (DDCI) Therapy in Early Idiopathic Parkinson's Disease Patients, With an Open-Label Extension
Brief Title: Early ParkinSon wIth L-DOPA/DDCI and OpicapoNe (EPSILON Study)
Acronym: EPSILON
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BIA-91067-303; 2020-005011-52 (EudraCT Number)
Record Dates: First submitted 2021-07-05; First posted 2021-07-27 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Parkinson
MeSH Terms: interventions — opicapone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Opicapone (Experimental): OPC will be taken orally once daily in the evening at least 1 hour after the last daily dose of L-DOPA/DDCI (considered the bedtime dose).
  Interventions: Drug: Opicapone 50 mg
- Matching placebo (Placebo Comparator): Matching placebo will be taken orally once daily in the evening at least 1 hour after the last daily dose of L-DOPA/DDCI (considered the bedtime dose).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Opicapone 50 mg — Capsule, 50 mg, Oral. Swallow whole with water, once daily at bedtime at least 1 hour after L-DOPA/DDCI
  Arms: Opicapone
Drug: Placebo — Capsule of to matching placebo, Oral. Swallow whole with water, once daily at bedtime at least 1 hour after L-DOPA/DDCI
  Arms: Matching placebo

SUMMARY:
Opicapone (OPC) is a third generation catechol O methyltransferase (COMT) inhibitor (COMTi) developed by BIAL-Portela & Cª, S.A. It is approved as adjunctive therapy to preparations of L-DOPA/DDCI in adult patients with Parkinson's disease and end-of-dose motor fluctuations who cannot be stabilized on those combinations. Carbidopa and benserazide are both DDCIs used in association with L DOPA. When OPC is co administered with L DOPA/DDCI, peripheral COMT is inhibited and thus L DOPA plasma levels increase, increasing L DOPA bioavailability. The purpose of this Phase III study is to explore the potential of OPC to enhance the clinical benefit of L-DOPA in L DOPA treated patients in the early stages of Parkinson's Disease (PD) (patients without end-of-dose motor fluctuations, 'non fluctuators').

DETAILED DESCRIPTION:
This is a Phase III study to evaluate the efficacy and safety of OPC in subjects with early idiopathic PD receiving treatment with L DOPA plus a DDCI, and who are without signs of any motor complication (consisting of fluctuations in the motor response and/or involuntary movements or dyskinesias).

After a screening period of up to 4 weeks, eligible subjects will be randomized into 1 of 2 treatment arms (OPC 50 mg, or placebo) in a 1:1 ratio, and enter a 24-week placebo-controlled, parallel-group, double blind period.

At the end of the double-blind period, subjects may enter an additional 1-year, open-label period, at the discretion of both the Investigator and subject, in which all subjects will be treated with OPC 50 mg.

A Post-study Visit (PSV) will be performed approximately 2 weeks after the End of Study Visit (EOS) or Early Discontinuation Visit (EDV).

Study treatment will be administered in combination with existing treatment of L-DOPA/DDCI.

ELIGIBILITY:
Inclusion Criteria:

1. Capable of giving signed informed consent.
2. Subjects must be 30 to 80 years of age, inclusive, at the time of signing the ICF.
3. Diagnosed with idiopathic PD according to the UK Parkinson's Disease Society Brain Bank Clinical Diagnostic Criteria within the previous 5 years.
4. Disease severity Stages 1 to 2.5 (according to the modified Hoehn & Yahr staging)
5. Signs of treatable motor disability for a minimum of 4 weeks before screening, with minimum threshold with MDS-UPDRS Part III score of ≥20 at both screening and Visit 2, despite stable anti-PD therapy (based on the investigator's judgment).
6. Receiving treatment with L-DOPA/DDCI (either controlled-release, immediate-release or combined controlled immediate-release) for at least 1 year, and at a stable regimen for at least 4 weeks prior to Visit 2 at a daily dose in the range 300 to 500 mg, 3 to 4 times a day.
7. Naive to COMT inhibitors (including OPC).
8. Male or female.

   • A male subject must agree to use contraception during the treatment period and until the PSV, and refrain from donating sperm during this period.

   • A female subject is eligible to participate if she is not pregnant , not breastfeeding, and at least 1 of the following conditions applies: i) Not a woman of childbearing potential (WOCBP) OR ii) A WOCBP who agrees to follow the contraceptive guidance during the treatment period and until the PSV.
9. Results of the screening laboratory tests are considered clinically acceptable by the Investigator (ie, not clinically relevant for the well-being of the subject or for the purpose of the study).

Exclusion Criteria:

1. Non-idiopathic PD (for example, atypical parkinsonism, secondary [acquired or symptomatic] parkinsonism, Parkinson-plus syndrome).
2. Signs of motor complications with a total score of MDS-UPDRS Part IV A+B+C greater than '0' (zero).
3. Treatment with prohibited medication: COMT inhibitors (eg, entacapone, tolcapone), antiemetics with antidopaminergic action (except domperidone) or Duopa™ (carbidopa/levodopa intestinal gel) within the 4 weeks before screening.
4. Concomitant use of monoamine oxidase (MAO-A and MAO-B) inhibitors (eg, phenelzine, tranylcypromine and moclobemide) other than those for the treatment of PD.
5. Previous or planned (during the entire study duration) deep brain stimulation.
6. Previous stereotactic surgery (eg, pallidotomy, thalamotomy) for PD or with planned stereotactic surgery during the study period.
7. Any investigational medicinal product within the 3 months (or within 5 half-lives, whichever is longer) before screening.
8. Any medical condition that might place the subject at increased risk or interfere with study assessments.
9. Past (within the past year) or present history of suicidal ideation or suicide attempts, as determined by a positive response ('Yes') to either Question 4 or Question 5 on the suicidal ideation portion of the Columbia-Suicide Severity Rating Scale (C-SSRS) (Screening questions)
10. Current or previous (within the past year) diagnosis of psychosis, severe major depression, or other psychiatric disorders that, based on the Investigator's judgment, might place the subject at increased risk or interfere with assessments.
11. A clinically relevant electrocardiogram (ECG) abnormality (relevance should be assessed by a cardiologist if needed).
12. Current evidence of unstable cardiovascular disease, including but not limited to uncontrolled hypertension, myocardial infarction with important systolic or diastolic dysfunction, unstable angina, congestive heart failure (New York Heart Association Class ≥III), and significant cardiac arrhythmia (Mobitz II 2nd or 3rd degree AV block or any other arrhythmia causing hemodynamic repercussions as symptomatic bradycardia or syncope).
13. Prior renal transplant or current renal dialysis.
14. Pheochromocytoma, paraganglioma or other catecholamine secretive neoplasm.
15. Known hypersensitivity to any ingredients of the study treatment.
16. History of neuroleptic malignant syndrome (NMS) or NMS-like syndromes, or non-traumatic rhabdomyolysis.
17. Malignancy within the past 5 years (eg, melanoma, prostate cancer), excluding cutaneous basal or squamous cell cancer resolved by excision.
18. Unstable active narrow-angle or unstable wide-angle glaucoma.
19. History of or current evidence of any relevant disease in the context of this study, ie, with respect to the safety of the subject or related to the study conditions, eg, which may influence the absorption or metabolism (such as a relevant liver disease) of the study treatment.
20. Any abnormality in the liver enzymes (alanine aminotransferase [ALT] and/or aspartate aminotransferase [AST]) >2 times the upper limit of the normal range, in the screening laboratory tests results.
21. Plasma sodium less than 130 mmol/L, white blood cell count less than 3000 cells/mm3, or any other relevant clinical laboratory abnormality that, in the Investigator's opinion, may compromise the subject's safety.
22. Positive SARS-CoV-2 test at screening.
23. Evidence of an ICD (one or more positive modules on the mMIDI)

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 410 (Actual)
Dates: Start 2021-05-31 (Actual); Primary Completion 2023-01-11 (Actual); Study Completion 2024-01-26 (Actual)

PRIMARY OUTCOMES:
Change from baseline (Visit 2) to the end of the double-blind period (Visit 9) in Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part III total score | Up to 24 weeks
  Double-Blind Period. Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part III questionnaire will be collected at visits 2, 3, 4, 6 and 9. MDS-UPDRS is a multimodal scale assessing impairment and disability consisting of 4 parts. Part III assesses the motor signs of PD and is rated by the investigator (score range 0-132). Part III contains 33 scores based on 18 items. A higher score indicates more severe symptoms of PD.
Change from open-label baseline (Visit 9) to the end of the open-label period (Visit 15) in MDS-UPDRS Part IV total score. | Up to 1-year.
  Open-Label Period. Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part IV questionnaire will be collected at Visits 9, 10, 11, 12, 13, 14 and 15. MDS-UPDRS is a multimodal scale assessing impairment and disability consisting of 4 parts. Part IV assesses the motor complications of PD, comprises 6 item (3 items for dyskinesia and 3 items for fluctuation; score range 0-24) and requires the physician to use historical and objective information to assess dyskinesia and motor fluctuations. A higher score indicates more severe symptoms of PD.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Centre "Asklepii", OOD, Dupnitsa, Bulgaria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: EU Clinical Trials Register — https://www.clinicaltrialsregister.eu/ctr-search/search?query=2020-005011-52
- See also: Movement Disorder Society - Unified Parkinson's Disease Rating Scale (MDS-UPDRS) — https://www.movementdisorders.org/MDS/MDS-Rating-Scales/MDS-Unified-Parkinsons-Disease-Rating-Scale-MDS-UPDRS.htm